CLINICAL TRIAL: NCT06977841
Title: Efficacy and Safety of Tegoprazan-Amoxicillin and Tegoprazan-Tetracycline Dual Therapy for Helicobacter Pylori Eradication: A Prospective, Randomized Controlled Study
Brief Title: Tegoprazan-Based Dual Therapy With Amoxicillin vs Tetracycline for H. Pylori Eradication
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Hospital (Xiamen), Fudan University (Other)
Responsible Party: Principal Investigator, Yucheng Zhu, Deputy Chief Physician, Zhongshan Hospital (Xiamen), Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYC-Hp2025
Record Dates: First submitted 2025-05-10; First posted 2025-05-18 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Helicobacter Pylori Eradication; High-dose Dual Therapy
MeSH Terms: interventions — tegoprazan; Amoxicillin; Capsules; Tetracycline; Bismuth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tegoprazan-Amoxicillin Dual Therapy (Experimental): Tegoprazan 50 mg orally twice daily (BID) before meals; Amoxicillin 750 mg orally four times daily (QID) after meals; Both administered for 14 consecutive days.
  Interventions: Drug: Tegoprazan; Drug: Amoxicillin 250Mg Cap
- Tegoprazan-Tetracycline Dual Therapy (Experimental): Tegoprazan 50 mg orally twice daily (BID) before meals; Tetracycline 500 mg orally four times daily (QID) after meals; Both administered for 14 consecutive days.
  Interventions: Drug: Tegoprazan; Drug: Tetracycline 500 Mg
- Tegoprazan-Amoxicillin-Tetracycline Triple Therapy (Active Comparator): Tegoprazan 50 mg orally twice daily (BID) before meals; Amoxicillin 1 g orally twice daily (BID) after meals; Tetracycline 500 mg orally three times daily (TID) after meals; All administered for 14 consecutive days.
  Interventions: Drug: Tegoprazan; Drug: Amoxicillin 250Mg Cap; Drug: Tetracycline 500 Mg
- Tegoprazan-Amoxicillin-Tetracycline-Bismuth Quadruple Therapy (Active Comparator): Tegoprazan 50 mg orally twice daily (BID) before meals; Amoxicillin 1 g orally twice daily (BID) after meals; Tetracycline 500 mg orally three times daily (TID) after meals; Bismuth agent (bismuth potassium citrate) 220 mg orally twice daily (BID) after meals; All administered for 14 consecutive days.
  Interventions: Drug: Tegoprazan; Drug: Amoxicillin 250Mg Cap; Drug: Tetracycline 500 Mg; Drug: Bismuth

INTERVENTIONS:
Drug: Tegoprazan — 50 mg twice daily (BID), d1-14, administered 30 minutes before morning and evening meals.
Drug: Amoxicillin 250Mg Cap — 750 mg four times daily (QID), d1-14, administered immediately after breakfast, lunch, dinner, and bedtime snack.
  Arms: Tegoprazan-Amoxicillin Dual Therapy; Tegoprazan-Amoxicillin-Tetracycline Triple Therapy; Tegoprazan-Amoxicillin-Tetracycline-Bismuth Quadruple Therapy
Drug: Tetracycline 500 Mg — 500 mg three times daily (TID), d1-14, postprandial after breakfast, lunch, and dinner.
  Arms: Tegoprazan-Amoxicillin-Tetracycline Triple Therapy; Tegoprazan-Amoxicillin-Tetracycline-Bismuth Quadruple Therapy; Tegoprazan-Tetracycline Dual Therapy
Drug: Bismuth — 220 mg BID, d1-14, administered 2-3 hours after tetracycline doses at lunch and dinner
  Arms: Tegoprazan-Amoxicillin-Tetracycline-Bismuth Quadruple Therapy

SUMMARY:
Current first-line Helicobacter pylori eradication protocols involve multidrug regimens comprising a proton pump inhibitor (PPI) or bismuth agent combined with dual antibiotics (e.g., clarithromycin, amoxicillin, quinolones, furazolidone, nitroimidazoles, or tetracycline) administered for 7-14 days. In China, the bismuth-containing quadruple therapy (BQT) remains the standard first-line treatment for H. pylori infection. However, BQT implementation is challenged by polypharmacy burdens, substantial adverse events, and suboptimal treatment adherence. Emerging evidence suggests that simplified dual therapies pairing acid suppressants (PPIs or potassium-competitive acid blockers [P-CABs]) with high-dose amoxicillin achieve comparable eradication rates to BQT while demonstrating superior tolerability and adherence profiles. Notably, the comparative efficacy of tetracycline-based versus amoxicillin-based dual regimens remains unexamined in controlled clinical trials. Our preliminary investigations established that optimized PPI-amoxicillin dual therapy achieves >90% eradication rates in treatment-naïve populations. Building on these findings, this prospective randomized controlled trial will comparatively assess the effectiveness of tegoprazan-a novel P-CAB exhibiting potent acid inhibition-when co-administered with either amoxicillin or tetracycline in H. pylori-positive adults. The investigation aims to establish an evidence framework for streamlining eradication protocols through pharmacodynamic optimization while mitigating antimicrobial resistance development.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) infection remains a significant global health burden, strongly associated with peptic ulcer disease, gastric cancer, and mucosa-associated lymphoid tissue (MALT) lymphoma. Current international and Chinese guidelines endorse multidrug regimens as first-line eradication therapy. The predominant approach, particularly in China, is bismuth-containing quadruple therapy (BQT). This regimen combines a proton pump inhibitor (PPI) or a bismuth agent with two antibiotics (selected from agents such as clarithromycin, amoxicillin, quinolones, furazolidone, nitroimidazoles, or tetracycline), typically administered for 7 to 14 days.

Despite its established position, BQT faces substantial challenges in real-world implementation. Polypharmacy, inherent in administering four distinct medications, creates a significant burden for patients, increasing the risk of dosing errors and non-adherence. Furthermore, the combination of multiple antimicrobials and bismuth frequently leads to substantial adverse events (e.g., gastrointestinal disturbances, taste alterations), which further compromise treatment adherence. Suboptimal adherence is a well-recognized factor contributing to treatment failure and the alarming rise in antimicrobial resistance (AMR).

In response to these challenges, simplified dual therapies have emerged as a promising alternative strategy. These regimens pair a potent acid suppressant - either a traditional PPI or the newer, more potent potassium-competitive acid blocker (P-CAB) class - with high-dose amoxicillin. Accumulating evidence suggests that such optimized dual therapies can achieve eradication rates comparable to BQT in treatment-naïve populations. Crucially, they demonstrate superior tolerability and significantly improved adherence profiles due to reduced pill burden and fewer side effects. This combination leverages the critical role of profound acid suppression in enhancing amoxicillin's efficacy against H. pylori while minimizing the use of additional antibiotics, thereby potentially mitigating AMR development.

However, a significant knowledge gap exists within this evolving paradigm. While amoxicillin-based dual therapy has been studied, the comparative efficacy of tetracycline-based dual therapy remains unexamined in rigorous controlled clinical trials. Tetracycline, a key component of some BQT regimens and salvage therapies, possesses distinct antimicrobial properties against H. pylori. Understanding its performance within a simplified dual therapy framework, particularly under potent acid suppression, is essential for expanding therapeutic options.

Building upon promising preliminary investigations demonstrating that optimized PPI-amoxicillin dual therapy consistently achieves >90% eradication rates in treatment-naïve patients, this research aims to further advance the field. We propose a prospective, randomized controlled trial to directly compare the effectiveness of two novel dual therapy regimens for first-line H. pylori eradication. Both regimens will utilize tegoprazan, a next-generation P-CAB known for its rapid, potent, and sustained acid-inhibitory effects. Tegoprazan will be co-administered with either high-dose amoxicillin or tetracycline.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 65 years;
2. H.pylori infection diagnosed by 13C-urea breath test;
3. The patient infected with Helicobacter pylori has never undergone eradication therapy.

Exclusion Criteria:

1. Allergy to any of the medications;
2. Zollinger-Ellison syndrome, GC, Upper gastrointestinal bleeding, or Active peptic ulcer;
3. Coexistence of significant concomitant illnesses, including heart disease, renal failure, hepatic disease, previous abdominal surgery, lactation, or pregnancy;
4. Patients who had used PPI/P-CAB drugs, and antibiotics in the past 12 weeks;
5. Unwillingness to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rate | 44 days
  Assessed by 13C-urea breath test (13C-UBT) at 30 days post-treatment. Eradication success was defined as a negative result (delta over baseline value <4‰).

SECONDARY OUTCOMES:
Frequency of the adverse events | 44 days
  Incidence rate of the adverse events, including dyspepsia, nausea, vomiting, abdominal pain, bloating, diarrhea, dizziness, headache, skin rash, fatigue and fever.
Compliance rate of the drugs | 44 days
  Compliance is defined as good when they had taken more than 80% of the total medication.

CONTACTS AND LOCATIONS:
Overall Officials: Yucheng Zhu, Ph.D., Principal Investigator — Zhongshan Hospital (Xiamen), Fudan University
Locations (1):
- Zhongshan Hospital (Xiamen), Fudan University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nan XP, Zhao HY, Guo LN, Zheng RQ, Wang XL, Wang YF, Su YH, Geng WR, Liu XL, Xu HM, Zhou KL, Guo YT, Cao JH, Han ZX, Kong QZ, Zuo XL, Li YQ, Li YY. Seven-Day Versus 14-Day Tegoprazan and Tetracycline-Containing Quadruple Therapy for First-Line Eradication of Helicobacter pylori Infection: A Randomized, Open-Label, Noninferiority Trial. Helicobacter. 2025 Mar-Apr;30(2):e70036. doi: 10.1111/hel.70036. PMID 40272011